CLINICAL TRIAL: NCT01433042
Title: Assessment the Performance of PillCam SB3 Capsule in Detecting Small Bowel Lesions in Patients
Brief Title: PillCam SB3 Capsule- Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD-304
Record Dates: First submitted 2011-09-07; First posted 2011-09-13 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2013-12

CONDITIONS: Small/Large Bowel
Keywords: small bowel disease
MeSH Terms: conditions — Cerebral Palsy | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capsule endoscopy (Experimental)
  Interventions: Device: capsule endoscopy

INTERVENTIONS:
Device: capsule endoscopy — capsule endoscopy procedure
  Other Names: CE

SUMMARY:
Study hypothesis: PillCam SB3 is a new capsule designed to provide an improved image quality, and improved SB and duodenum tissue coverage due to Adaptive Frame Rate (AFR) of 2-6 fps, which will create more images for evaluation, and therefore should improve diagnostic accuracy.

Proposed Design: to enroll up to 230 patients with symptoms suggesting the presence of small bowel disease.

Preparation for procedure will include 12 hours fasting prior to the capsule ingestion

Patients will undergo a standard capsule endoscopy. Patients will be allowed to drink clear liquids 2 hours post ingestion, and eat 4 hours post ingestion.

Diagnostic yield of the SB3 will be calculated The Physician's subjective assessment of capsule performance will be captured

DETAILED DESCRIPTION:
* Purpose of study- To assess the performance of PillCam SB3 capsule in detecting small bowel lesions in patients
* Study design- Feasibility study
* Number of subjects- Up to 200
* Subject population- Patients with symptoms suggestive of small bowel disease and whom are eligible and indicated for SB capsule endoscopy
* No of centers- 4
* Duration of enrollment up to 12 months from IRB approval to enroll study patients
* Duration of follow-up 1 week after capsule procedure.
* Primary objectives To evaluate the performance of SB-3 system in patients as per physician questionnaire

ELIGIBILITY:
Inclusion criteria:

1. Patient age is ≥ 18 years old,
2. Patients with history suggestive and /OR symptoms suggestive of small bowel disease and whom are eligible and indicated for SB capsule endoscopy,
3. Patient and/or legal guardian is able and agrees to sign the Informed Consent Form

Exclusion criteria

1. Patient has dysphagia,
2. Patient is known or is suspected to suffer from intestinal obstruction,
3. Patient has known previous stricture/obstruction of the SB or colon,
4. Patient has a cardiac pacemakers or other implanted electro medical devices, 5. Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child-bearing potential and do not practice medically acceptable methods of contraception,

6. Patient is expected to undergo MRI examination within 7 days after ingestion of the capsule, 7. Patient has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator, 8. Patient has any condition, which precludes compliance with study and/or device instructions, 9. Patient suffers from life threatening conditions, 10. Patient is currently participating in another clinical study, 11. Patient has known slow gastric emptying time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Adler, Prof, Principal Investigator — Medtronic - MITG
Locations (4):
- Bikur Holim medical center, Jerusalem, Israel
- University Hospital, Bucharest, Romania
- Servicio de Digestivo Hospital de Navarra, Pamplona, Spain
- Skane University Hospital, Lund University, Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients enrolled in this study were indicated to undergo SB capsule endoscopy and/or had symptoms suggestive of SB disease. 225 patients were enrolled in this study recruitment period: August 2011 till September 2012. recruitment performed at Gastroenterlogy clinics and departments
Pre-assignment Details: After obtaining the consent, subjects were assessed for eligibility to participate based on the eligibillity criteria. Each patient underwent a PillCam SB3 procedure. Preparation for the procedure included a 12 hours fast prior to the PillCam SB3ingestion.
  Patients were allowed to drink clear liquids 2 hours and eat 4 hours post ingestion.
Groups:
- Capsule Endoscopy: capsule endoscopy : capsule endoscopy procedure
Period: Overall Study
Arm/Group | Capsule Endoscopy
Started | 225
Completed | 224
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: 18 years and older patients with history suggestive and /or symptoms suggestive of small bowel disease and whom are eligible and indicated for SB capsule endoscopy and agreed to sign ICF
Arm/Group | Capsule Endoscopy
Number analyzed (Participants) | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 157
  >=65 years | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 113
Region of Enrollment [Number; unit: participants]
  Spain | 66
  Romania | 19
  Israel | 76
  Sweden | 64

OUTCOME MEASURES:

1. Primary Outcome: Precentage of SB3 Images That Were Graded as Superior in Image Quality to SB2 by the Physicians
Description: precentage of SB3 images that were graded as superior in image quality to SB2 by the physicians
Time Frame: up to 6 months from end of recruitment
Population: Five (2%) cases were excluded from the efficacy analysis due to the following :
  * 1 patient withdrawn prior to any procedure.
  * 1 patient did not meet the inclusion criteria
  * 3 cases, the capsule remained in the stomach during the entire procedure.
  Therefore, 220 cases are included in the efficacy analysis.
Measure: Number; unit: percentage of cases
Arm/Group | Capsule Endoscopy
Number analyzed (Participants) | 220
percentage of cases | 98
Statistical Analysis 1: Comparison: Capsule Endoscopy; Primary Endpoint o Physician's subjective assessment questionnaire was evaluated in a quality manner. The physicians were required to assess the performance of SB3 system as compare to SB2 by answering a short questionnaire. The physicians were requested to indicate whether capsule SB3 was better as compared to SB2; Test type: Superiority or Other; percentage — since the study results analysis is purley discriptive no P value and confidence interval was used for the analysis; percentage of SB3 images graded as superior in image quality to SB2; percentage = 98 — since the study results analysis is purley discriptive no P value and confidence interval was used for the analysis

ADVERSE EVENTS:
Time Frame: two weeks after capsule procedure
Arm/Group | Capsule Endoscopy
Serious Adverse Events (participants affected / at risk) | 1/225
Other Adverse Events (participants affected / at risk) | 0/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capsule Endoscopy (N=225)
Serious Cardiovascular event (Cardiac disorders) | 1 (1) — One serious Cardiovascular adverseevent -not related to capsule procedure was reported within this study: the patient died one day after capsule procedure as a result of cardiovascular event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days